CLINICAL TRIAL: NCT01130376
Title: A Randomised, Open Labelled, Phase I, Safety, Toxicity, and Exploratory Immunogenicity Evaluation of Therapeutic Immunisation +/- IL-2, GM-CSF and Growth Hormone in HIV-1 Infected Subjects Receiving Highly Active Anti-retroviral Therapy
Brief Title: Novel Interventions in HIV-1 Infection
Acronym: IMIRC1003
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Data from the 12 patients recruited has now been analysed, and it has been determined that it is sufficient to meet the study objectives.
Sponsor: Imperial College London (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRO930; G0501957 (Other Grant/Funding Number: Medical Research Council UK); 2008-000575024 (Registry Identifier: EudraCT)
Record Dates: First submitted 2010-05-25; First posted 2010-05-26 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2012-09

CONDITIONS: HIV-1 Infection
Keywords: Immune based therapy; Therapeutic vaccination; cytokine therapy; HIV therapeutic vaccine
MeSH Terms: interventions — Interleukin-2; aldesleukin; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Vaccine and cytokines (Experimental): Day 0: Patients receive GTU-MultiHIV B clade vaccine 1mg/ml administered as 10 intradermal injections of 100 µl/injection.
  Day 7-11: One week following this, patients receive a 5 day course of Cytokines: Aldesleukin (IL-2) Novartis UK (BD; 8 hours apart) 5 million units administered by SC injection. Sargramostim (GM-CSF) - Leukine™, Berlex Seattle US 150ug SC once daily 4 hours from rhIL-2 injections.
  Day 14-18: The following week, patients rhGH (Saizen™, Serono International, Geneva, Switzerland) 4mg/day self-administered SC.
  Further vaccine boosters are given on day 42 and day 84. GTU-MultiHIV B clade vaccine 1mg/ml being administered as 10 intradermal injections of 100 µl/injection.
  Interventions: Biological: GTU-MultiHIV B clade vaccine1mg; Drug: Interleukin-2; Drug: GM-CSF; Drug: Growth Hormone
- Vaccine alone (Active Comparator): Day 0: Patients are given GTU-MultiHIV B clade vaccine 1mg/ml administered as 10 intradermal injections of 100 µl/injections.
  Day 42: GTU-MultiHIV B clade vaccine as day 0.
  Day 84: GTU-MultiHIV B clade vaccine as day 0.
  Interventions: Biological: GTU-MultiHIV B clade vaccine1mg
- Cytokines alone (Active Comparator): Day 7-11: One week following this, patients receive a 5 day course of Cytokines: Aldesleukin (IL-2) Novartis UK (BD; 8 hours apart) 5 million units administered by SC injection. Sargramostim (GM-CSF) - Leukine™, Berlex Seattle US 150ug SC once daily 4 hours from rhIL-2 injections.
  Day 14-18: The following week, patients rhGH (Saizen™, Serono International, Geneva, Switzerland) 4mg/day self-administered SC.
  Interventions: Drug: Interleukin-2; Drug: GM-CSF; Drug: Growth Hormone

INTERVENTIONS:
Biological: GTU-MultiHIV B clade vaccine1mg — Dose given is 1mg/ml administered as 10 intradermal injections of 100 µl/injection distributed as 5 intradermal injections /left and right arm
  Arms: Vaccine alone; Vaccine and cytokines
Drug: Interleukin-2 — 5 Million Units administered twice daily for 5 days by subcutaneous injection on days 7, 8, 9, 10, and 11 after first vaccination. .
  Other Names: Aldesleukin; Proleukin
  Arms: Cytokines alone; Vaccine and cytokines
Drug: GM-CSF — 150 ug administered subcutaneously once daily 4 hours from IL-2 injections
  Other Names: Sargramostim; Leukine
  Arms: Cytokines alone; Vaccine and cytokines
Drug: Growth Hormone — 4mg/day will be self administered by Subcutaneous injection for 5 days on days 14, 15, 16, 17 and 18 following first vaccination
  Other Names: Serono International, Geneva, Switzerland
  Arms: Cytokines alone; Vaccine and cytokines

SUMMARY:
For several years there has been interest in why some people with HIV-1 progress more slowly to disease and have longer survival without Highly Active Antiretroviral Therapy (HAART) than others. The investigators and others have identified a few HIV positive individuals who can control their viral load for many years without HAART, these rare individuals do not lose their HIV-1-specific cellular immune responses, which are very important for controlling viral load. This group is referred to as long-term non-progressors (LTNP). Unlike LTNP the majority of HIV-1 infected individuals are chronic progressors (CP) who do not make effective HIV-1-specific cellular immune responses, even when on HAART. We propose to use a novel DNA vaccine boosted with immune based therapy (cytokines and hormones) to try to regenerate the missing HIV-1-specific cellular immune responses to make chronically infected HIV-1+ persons more like LTNP.

By injecting this novel DNA vaccine and immune based therapy into the people who are already infected with HIV-1, the immune system may be stimulated to mount a greater immune response not only to the vaccines but also to real HIV-1 particles and HIV-1-infected cells.

DETAILED DESCRIPTION:
This will be a randomised, Phase I, open label comparative study running for 52 weeks (2 screen visits 2 weeks apart followed by 48 weeks of study). 50 patients will be screened in the initial phase of which 30 clade B infected individuals will be randomised into the study, which will consist of 3 arms:

Arm 1 will ascertain vaccine safety and toxicity in the presence of cytokine/hormone therapy.

Arm 2 will identify vaccine safety and toxicity.

Arm 3 will indicate safety and toxicity of cytokine/hormone therapy.

The target patients are chronically HIV-1 clade B infected persons who will have had a nadir CD4 T-cell count of >200 cells/ul blood before they started ART. The current CD4 T-cell count should be >400 cells/ul blood. Patients may have received ART for any length of time, but currently should be receiving NNRTI or boosted-PI based HAART, and have a viral load below the level of detection (50 copies/ml plasma). Patients will be bled on two occasions before commencing IBT regimens, in order to establish baselines, and then at regular intervals thereafter (weeks 0,1,2,4,6,8,12,16,24 and 48).

The treatment regimens are consistent with previous findings in animal models which suggest that administration of IL-2 during the antigen-specific T-cell contraction phase of an immune response (between 8 and 15 days post-vaccination) may preserve and lengthen clinically relevant responses. Furthermore studies in man have demonstrated that IL-2 administered before immunisation in ART-treated HIV-1-infected patients does not increase specific lymphoproliferation of T cells.

Recent preliminary studies in HIV-1-infected individuals using tetanus vaccines the investigators have shown that IL-2 administered after immunisation may be more effective at inducing sustained tetanus-specific responses than IL-2 administered before immunisation or together with immunisation. The dosages used in this study are based on those used in previous pilot studies of the administration of IL-2 + GM-CSF and rhGH and at these levels the drugs have been shown to have both positive effect on the immune response and demonstrated clinical benefit whilst being at a level which is safe and well tolerated in HIV-1 positive individuals. The dosage of the vaccine was based on a previous study where a dosage of this level has been shown to induce an immune response although this response was transient. In summary the investigators aim to increase the survival of vaccine responses through the administration of cytokines/hormones and boost memory responses with further rounds of immunisation.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV-1 positive result.
* Stable on HAART.
* Two screening viral loads of <50 cps/ml on 2 consecutive occasions at least one month apart.
* CD4 T cell count of >400 cells/ul.
* Nadir CD4 T cell count of >200 cells/ul.
* Over 18 years of age.
* Willing and able to provide informed consent.
* Female subjects must not be pregnant or lactating.
* Subjects must be using adequate double barrier method of contraception as appropriate.

Exclusion Criteria:

* Prior therapeutic vaccination.
* Acute illness within 2 weeks of the start of the study.
* Prior immunomodulatory therapy (e.g. IL-2, rhGH, GCSF, GM-CSF, HU)
* Receiving immunosuppressive medication (e.g. Steroids)
* Participation in other vaccine trials currently
* Patients with diabetes mellitus type 2
* Patients with cardiac abnormalities
* Patients with pre-existing autoimmune disease
* Patients with active neoplasia
* Patients with evidence of any progression or recurrence of an underlying intra-cranial lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be analysis of safety and toxicity data in relation to grade 3 or above laboratory or clinical serious adverse event (SAE) which can be attributed to the treatments given | Weekly

SECONDARY OUTCOMES:
The secondary immunological outcomes will be percentage change from baseline to study time point in defined cellular immune responses. | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Nesrina Imami, MD/PhD, Principal Investigator — Imperial College London
Locations (1):
- St. Stephen's AIDS Trust, London, United Kingdom

REFERENCES:
- [Derived] Herasimtschuk A, Downey J, Nelson M, Moyle G, Mandalia S, Sikut R, Adojaan M, Stanescu I, Gotch F, Imami N. Therapeutic immunisation plus cytokine and hormone therapy improves CD4 T-cell counts, restores anti-HIV-1 responses and reduces immune activation in treated chronic HIV-1 infection. Vaccine. 2014 Dec 5;32(51):7005-7013. doi: 10.1016/j.vaccine.2014.09.072. Epub 2014 Oct 22. PMID 25454870
- See also: research team web page — http://www1.imperial.ac.uk/departmentofmedicine/divisions/infectiousdiseases/immuno/candw/immreconhiv/